CLINICAL TRIAL: NCT07139782
Title: Home-Based Photo-Biomodulation for Management of Lymphoedema and Radiation Fibrosis in Patients After Head and Neck Cancer: A Single-Arm Feasibility Trial
Acronym: HOME-PBM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 115976
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; photo-biomodulation; radiation fibrosis; lymphoedema; physiotherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Fibrosis Syndrome; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): RIANCORP
  1. The therapist will complete 5 minutes of manual lymphatic drainage (MLD) prior to photo-biomodulation (PBM)
  2. The therapist will apply the device for 60 secs each at 14 - 25 points on the face and neck. Most patients will need application of the device at 15 to 20 points The Riancorp runs for 60 seconds, providing 1.5 j/cm2 in 60 seconds. The Riancorp has an in-built timer that signals the end of 60 seconds.
  HANDYCURE PROTOCOL The Handycure device will be used at home by the patients, in addition to the usual care. Education, including written instruction sheets in how patients are to perform MLD, and use of the device will be provided.
  The device is to be used once/day on the prescribed days (Wks 1-6 3x/wk; Wks 7-10 x2/wk; Wks 11-12 x1/wk)
  1. Patients will complete 5 min of MLD prior to PBM
  2. They will then apply the device for 5 minutes at each point.
  Telehealth physio (wks 1, 6 and 9) post baseline will check usage, adherence and monitor safety.
  Interventions: Device: Riancorp LTU-904 Laser and Handycure® (Medical Quant)

INTERVENTIONS:
Device: Riancorp LTU-904 Laser and Handycure® (Medical Quant) — Riancorp: At the first intervention session the therapist will apply the device for 60 secs each at 14 - 25 points on the face and neck. Most patients will need application of the device at 15 to 20 points The Riancorp runs for 60 seconds, providing 1.5 j/cm2 in 60 seconds.
  Handycure: used by patients at home once/day on the prescribed days (Wks 1-6 3x/wk; Wks 7-10 x2/wk; Wks 11-12 x1/wk) 1. Patients will apply the device for 5 minutes at each point as instructed by the physiotherapist.

SUMMARY:
This feasibility trial will test the use of photo-biomodulation (PBM) therapy, predominantly self-delivered in the patient's home for 12-weeks, following completion of radiotherapy treatment for head and neck cancer.

The primary objective is to establish feasibility of recruitment (uptake). Secondary objectives are to assess safety, additional elements of feasibility (adherence to the intervention, return of the device and attrition at the 3-month follow-up appointment) and acceptability of the trial to patients.

Secondary measures will be performed to assess trends in effects of the intervention (pre-post intervention, within-group measures) for managing lymphoedema and radiation fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has provided written informed consent using the HOME-PBM patient information and consent form
2. Patient is referred to the Lymphoedema Clinic for the management of head and neck lymphoedema and/or radiation fibrosis
3. Previously received curative-intent treatment (surgery and/or [chemo]radiotherapy) for mucosal head and neck cancer
4. Patient is able to attend appointments in person
5. Adults aged 18 years or older at Screening
6. Patient able to speak and read English

Exclusion Criteria:

1. Patient has cognitive impairment that in the opinion of the Investigator would interfere with their ability to participate in the trial (e.g., complete outcome measures, perform the intervention)
2. Residual or recurrent disease within the head and neck
3. Has a diagnosis of photosensitive disorder (cutaneous porphyria, xeroderma pigmentosum, etc.)
4. Patient has tuberculosis or another form of virulent bacteria
5. Patient has a contraindication to receiving PBM treatment
6. Patient has no internet enabled device for telehealth video follow-up appointment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-04 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Uptake (trial consent rate) | Throughout the trial for 12-months of recruitment
  Consent rate and reasons for declining trial participation

SECONDARY OUTCOMES:
Adverse events | Throughout the trial for 12-months of recruitment
  Safety will be measured by the number of adverse events (AEs) related to the trial intervention and outcome assessments and reported according to the Common Terminology Criteria for Adverse Events version 5.
Acceptability | Three months post baseline
  Assessed by inviting a subgroup of patients (n=15-20) to complete an individual semi-structured interview by telephone or videoconferencing.
Program adherence | Throughout the trial for 12-months of recruitment and completion of 3-month follow-up
  The number of scheduled clinic and telehealth sessions attended
Program adherence | Throughout the trial for 12-months of recruitment and completion of 3-month follow-up
  Adherence to prescribed unsupervised intervention (PBM) sessions
Retention | 3-months post-baseline
  Patient retention at the follow-up assessment
Neck circumference | Baseline and 3-months post-baseline
  Neck circumference to be measured using the Assessment of Lymphoedema of the Head and Neck (ALOHA) method
Lymphoedema | Baseline and 3-months post-baseline
  The MD Anderson Cancer Centre Head and Neck Lymphoedema (MDACC HNL) Rating Scale will be used by the therapist to rate the degree of lymphoedema
Percentage water content (PWC) of skin | Baseline and 3-months post-baseline
  Percentage water content of the skin to be performed using the Lymph Scanner
Cervical spine range of motion | Baseline and 3-months post-baseline
  Neck range of motion to be measured with a digital goniometer
Shoulder range of motion | Baseline and 3-months post-baseline
  Shoulder range of movement to be measured with a digital goniometer
Trismus | Baseline and 3-months post-baseline
  Maximal incisal opening (trismus): The distance (in millimetres) between the edges of the maxillary and mandibular central incisors will be measured using the Therabite Range of Motion Scale.
Health-related quality of life | Baseline and 3-months post-baseline
  EORTC QLQ-HN43

CONTACTS AND LOCATIONS:
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided